CLINICAL TRIAL: NCT03171207
Title: Evaluation of a Novel Gait Training Device Using a Pressurized Lower Body Suit to Support Body Weight
Brief Title: Evaluation of a Novel Gait Training Device to Support Body Weight
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lite Run Inc. (Industry)
Collaborators: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency); TREAT (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4698-A
Record Dates: First submitted 2017-05-24; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Stroke; Brain Injuries, Traumatic; Spinal Cord Injuries; Gait Disorders, Neurologic
Keywords: Gait Therapy
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Spinal Cord Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Start with Lite Run Gait Trainer (Experimental): Patients start therapy with the Lite Run Gait Trainer device, followed by a Current Harness System in an ABAB design.
  Interventions: Device: Lite Run Gait Trainer; Device: Current Harness System
- Start with Current Harness System (Experimental): Patients start therapy with a Current Harness System, followed by the Lite Run Gait Trainer in an ABAB design.
  Interventions: Device: Lite Run Gait Trainer; Device: Current Harness System

INTERVENTIONS:
Device: Lite Run Gait Trainer — The Lite Run Gait Trainer is a novel device with pneumatic pants that can be used to assist with body support assisted gait therapy.
Device: Current Harness System — There are a variety of harness systems (e.g., ceiling lift, Lite Gait) that are currently used to assist with body support assisted gait therapy.

SUMMARY:
A novel body weight support device that uses pressurized pants may provide advantages in delivering gait therapy. The objectives of this study are to test the following hypotheses that 1) the novel device will allow for increased body weight support while improving or maintaining the same level of patient comfort; 2) the novel device will yield greater patient satisfaction with gait therapy relative to current harness systems; 3) therapists will be more satisfied with the use of the novel device relative to current harness systems; 4) the use of the novel device will require less total therapist time than a harness comparator; 5) the use of the novel device will increase therapeutic treatment time when compared with current harness systems.

DETAILED DESCRIPTION:
This is a single group repeated measures ABAB design. The study will include four sessions for each participant, with two sessions conducted using a novel Lite Run Gait Trainer device (Lite Run, Inc., Minneapolis, MN) and two sessions conducted using the comparator method of choice by the physical therapist (harness system). The initial condition (harness or Lite Run) will be randomized. The overall gait training physical therapy session will follow standard of care; the only factor that will change will be the assistive device used during therapy (harness or Lite Run).

Participants will include 10 VA inpatients receiving physical therapy at the Minneapolis VA Health Care System (MVAHCS). Patients will be recruited from three VA rehabilitation units: Physical Medicine and Rehabilitation (PM&R), Spinal Cord Injury and Disease (SCI/D) Center, and Community Living Center (CLC). Participants will have a range of diagnoses: stroke, traumatic brain injury, spinal cord injury, wounds, obesity.

The number of therapists and their time involvement will be tracked as a primary outcome measure in this study. The effectiveness of treatment will also be assessed for both assistive device methods. The total amount of therapeutic treatment time will be measured as the time spent by the patient in an upright position. At the end of each therapy session, participants will also be asked to rate their pain (comfort), perceived level of exertion, and will fill out a questionnaire about their experience with the Lite Run Gait Trainer. The physical therapists involved in the study will also provide their feedback.

ELIGIBILITY:
Inclusion Criteria:

* Veterans age: 18-90 years, male or female,
* Who are receiving physical therapy as an inpatient at MVAHCS,
* Have Functional Independence Measure (FIM) scores of 0 or 1 (out of 7) in at least one of the five domains of motor tasks: 1) bed, chair, and wheelchair transfers, 2) toilet transfers, 3) tub/shower transfers, 4) walk/wheelchair locomotion, 5) stair locomotion,
* Who are determined by VA standards to require at least 35 pounds of physical support, such that 2 or more physical therapists and/or aides are needed during therapy, and
* Are able to understand informed consent.

Exclusion Criteria:

* Patients who have active clostridium difficile,
* An acute diagnosis of deep vein thrombosis, chronic deep vein thrombosis, or phlebitis (unless cleared by clinician to participate in the study),
* A lower body pressure ulcer worse than grade one (EPUAP), or an open wound,
* A history of any drug-resistant pathogen, such as Methicillin-resistant Staphylococcus aureus (MRSA) or Vancomycin-resistant enterococci (VRE), ESBL producing gram-negative bacilli, or others,
* Weigh more than 350 lbs.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of therapists and/or aides required for a therapy session | From beginning of each therapy session to the end of each therapy session (approximately 60 minutes)
  Count of therapists and/or aides involved in therapy
Total therapist and/or aide time involved in a session | From beginning of each therapy session to the end of each therapy session (approximately 60 minutes)
  Total cumulative time (min) for all therapists and aides involved in a therapy session

SECONDARY OUTCOMES:
Total time spent by patient in an upright position during a therapy session | From beginning of each therapy session to the end of each therapy session (approximately 60 minutes)
  Total time spent (min) by patient in an upright position
Amount of unweighting | Will be assessed during the first five minutes of each therapy session following fitting of harnessing system
  The amount of unweighting (pounds of body support) will be measured using a scale
Numerical pain rating scale | Will be assessed at the end of each therapy session (approximately 60 minutes)
  Patient rating of pain (on a 0-10 numerical scale) will be assessed at the end of each therapy session
Patient Satisfaction | Will be assessed after the last session in each study arm (i.e., after two therapy sessions lasting approximately 60 minutes each)
  The first 8 questions of the Modified Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) will be given
Therapist Satisfaction | Will be assessed at the end of the study (i.e., after four therapy sessions lasting approximately 60 minutes each)
  The first 8 questions of the Modified Quebec User Evaluation of Satisfaction with assistive Technology (QUEST) will be given

CONTACTS AND LOCATIONS:
Overall Officials: Sara R Koehler-McNicholas, PhD, Principal Investigator — Minneapolis Veterans Affairs Medical Center

IPD SHARING:
Plan to Share IPD: No